CLINICAL TRIAL: NCT06713889
Title: Identifying Biological Markers of Cardiovascular Events in Patients With Aortic Stenosis or TAVI
Acronym: Bio-TAVI
Status: Recruiting | Type: Observational
Sponsor: Hospices Civils de Lyon (Other)
Responsible Party: Sponsor
Other Study IDs: 69HCL21_1209; 2024-A01552-45 (Other: ID-RCB)
Record Dates: First submitted 2024-11-27; First posted 2024-12-03 (Actual); Last update posted 2025-11-25 (Actual); Status verified 2025-10

CONDITIONS: Aortic Stenosis
Keywords: Aortic stenosis; TAVI; Cardiology; Biomarkers
MeSH Terms: conditions — Aortic Valve Stenosis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — In order to build up the cohort's biocollection (serotheque, plasmatheque), additional tubes will be taken at the same time as routine blood sampling. At each sampling time, 2 dry tubes of 4 ml, 1 EDTA tube of 4 ml, and 1 heparinised tube of 4 ml, i.e. a total of 16 ml per sampling time.
  Group A patients will be sampled at inclusion, before, during and after the TAVI procedure, at 1 month follow-up and at 1 year follow-up, for a total of 120 ml. Patients in groups B and C will be sampled at inclusion, 1 month follow-up, 1 year follow-up and 2 years follow-up, for a total of 80 ml.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- Group A: Patients with symptomatic severe aortic stenosis, with indication for TAVI. They are followed at inclusion, during hospitalisation of the TAVI procedure, at 1-month follow-up, at 1-year follow-up and by phone at 2 years follow-up.
  Interventions: Biological: Biocollection; Behavioral: Quality of life questionnaires
- Group B: Patients with asymptomatic severe aortic stenosis, without indication for TAVI. They are followed at inclusion, at 1-month follow-up, at 1-year follow-up and at 2 years follow-up.
  Interventions: Biological: Biocollection; Behavioral: Quality of life questionnaires
- Group C: Patients with asymptomatic middle aortic stenosis, without indication for TAVI. They are followed at inclusion, at 1-month follow-up, at 1-year follow-up and at 2 years follow-up.
  Interventions: Biological: Biocollection; Behavioral: Quality of life questionnaires

INTERVENTIONS:
Biological: Biocollection — At each sampling time, 2 dry tubes of 4 ml, 1 EDTA tube of 4 ml, and 1 heparinised tube of 4 ml, i.e. a total of 16 ml per sampling time.
  Group A patients will be sampled at inclusion, before, during and after the TAVI procedure, at 1 month follow-up and at 1 year follow-up, for a total of 120 ml. Patients in groups B and C will be sampled at inclusion, 1 month follow-up, 1 year follow-up and 2 years follow-up, for a total of 80 ml.
Behavioral: Quality of life questionnaires — EQ-5D-5L and HAD questionnaire at inclusion, 1 month follow-up, 1 year follow-up and 2 years follow-up

SUMMARY:
Aortic stenosis, a common cardiovascular disease, is pathophysiologically associated with a chronic inflammatory myocardial reaction and fibrosis leading to cardiac dysfunction and impaired coronary perfusion. These elements may precede the onset of symptoms. The assessment of inflammatory and fibrosis factors (in particular by means of biomarkers) in patients with aortic stenosis will make it possible to identify asymptomatic patients at greater risk who could benefit from intervention earlier. This is part of a personalised medicine adapted to the patient.

Patients will be recruited during their TAVI (Transcatheter Aortic Valve Implantation) assessment consultation. If the patient agrees to take part in the study, information relating to routine care procedures will be collected (patient history, clinical examinations, electrocardiogram, echography, coronary angiography, TAVI procedure if applicable, biology).

Outside of routine care, a biocollection will be established (serum, plasma), quality of life questionnaires will be carried out and adverse events will be collected where present.

Patients will be divided into 3 groups according to the indication for TAVI (Group A - symptomatic severe aortic stenosis with indication for TAVI, Group B - asymptomatic severe aortic stenosis without indication for TAVI, Group C - asymptomatic moderate aortic stenosis without indication for TAVI).

The main objective is to compare the levels of biomarkers of inflammation and fibrosis between the 3 groups at each sampling time common to all three groups between inclusion and 1-year follow-up.

ELIGIBILITY:
Inclusion Criteria:

* Patients >=18 years of age
* Patient with symptomatic or asymptomatic severe or moderately severe aortic stenosis (according to the recommendations of the European Society of Cardiology - ESC).
* No opposition.

Exclusion Criteria:

* Conjunctive heart disease (e.g. amyloidosis).
* Presence of a contraindication to TAVI.
* Impossibility of giving the subject informed information.
* Privation of civil rights (curatorship, tutorship, protection of justice).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: 125 patients will be selected from among those seen in consultation for aortic stenosis assessment in the cardiology departments of the Louis Pradel and Croix-Rousse hospitals.
Sampling Method: Non-Probability Sample
Enrollment: 125 (Estimated)
Dates: Start 2024-12-19 (Actual); Primary Completion 2027-06 (Estimated); Study Completion 2028-06 (Estimated)

PRIMARY OUTCOMES:
Comparing biomarkers | At V0 (inclusion), V4 (1-month follow up) and V5 (1-year follow up).
  The primary endpoint is the level of biomarkers of inflammation and fibrosis in the 3 groups of patients.

CONTACTS AND LOCATIONS:
Overall Officials: Ahmad HAYEK, MD, Principal Investigator — Plateau technique interventionnel - Hôpital Louis Pradel, GHE
Locations (2):
- France (2):
  - Hospices Civils de Lyon - Hôpital Croix Rousse, Lyon
  - Hospices Civils de Lyon - Hôpital Louis Pradel, Lyon